CLINICAL TRIAL: NCT03427749
Title: Multi-Center Evaluation of Feasibility of SPECT Measurement of Myocardial Blood Flow and Reserve
Status: Completed | Type: Observational
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 20170797
Record Dates: First submitted 2018-02-02; First posted 2018-02-09 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease
Keywords: Myocardial Blood Flow; SPECT
MeSH Terms: conditions — Coronary Artery Disease | interventions — Tomography, Emission-Computed, Single-Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SPECT Imaging with 99mTc-Tetrofosmin: Patients will be recruited from those referred to the local site's Diagnostic Imaging Department for SPECT myocardial perfusion imaging (MPI) and who have an intermediate to high pre-test likelihood of disease (Diamond-Forrester criteria ≥ 30%). Research imaging will consist of a SPECT acquisition at the time of rest and stress radiotracer injection in addition to the standard (delayed) clinical stress/rest SPECT scan with 99mTc-tetrofosmin
  Interventions: Diagnostic Test: SPECT Imaging with 99mTc-Tetrofosmin Research Imaging

INTERVENTIONS:
Diagnostic Test: SPECT Imaging with 99mTc-Tetrofosmin Research Imaging — This is an observational study; patients will be managed according to the standard clinical care of the local site. Study end will be defined as completion of all SPECT imaging at rest and stress. Studies will be acquired at 6 initial sites with mixed prior experience at MBF imaging, to demonstrate feasibility of use in a clinical setting.

SUMMARY:
Patients will be recruited from those referred to the local site's Diagnostic Imaging Department for SPECT myocardial perfusion imaging (MPI) ,who have an intermediate to high pre-test likelihood of disease (Diamond-Forrester criteria ≥ 30%) and are clinically indicated to have an MBF study.

DETAILED DESCRIPTION:
Patients will be recruited from those referred to the local site's Diagnostic Imaging Department for SPECT myocardial perfusion imaging (MPI), who have an intermediate to high pre-test likelihood of disease (Diamond-Forrester criteria ≥ 30%) and are clinically indicated to have an MBF study. Research imaging will consist of a SPECT acquisition at the time of rest and stress radiotracer injection in addition to the standard (delayed) clinical stress/rest SPECT scan with 99mTc-tetrofosmin. This is an observational study; patients will be managed according to the standard clinical care of the local site. Where available, a CT scan will also be acquired for attenuation and/or scatter correction. Studies may be one day (rest/stress or stress/rest) or two day (rest and stress on separate days) All studies will be analyzed locally but the raw data will also be anonymized and forwarded to the core facility for reprocessing. Central processing will allow comparison between sites and the repeat processing will provide an estimate of inter-operator variability in the measurements. The core lab will also compare the relative perfusion from immediate and delayed imaging for image quality and diagnostic accuracy (visual and quantitative).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* BMI ≤ 40 kg/m2
* Able and willing to comply with the study procedures
* Written informed consent
* Intermediate to high probability of CAD
* Suspected or known CAD on a stable medication regime

Exclusion Criteria:

* History or risk of severe bradycardia (heart rate < 50 beats per minute) not related to chronotropic drugs
* Known second- or third-degree AV block without pacemaker
* Dyspnea (NYHA III/IV), wheezing asthma or COPD
* Coronary artery bypass graft (CABG) surgery within 60 days prior to screening or within 45 days after consent (early revascularization)
* Percutaneous coronary intervention (PCI) within 30 days prior to screening or within 45 days following consent (early revascularization)
* Recent use of dipyridamole, dipyridamole-containing medications (e.g. Aggrenox)
* Known hypersensitivity to dipyridamole or adenosine
* Breastfeeding or pregnancy
* Claustrophobia or inability to lie still in a supine position
* Unwillingness or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be adult male and female patients who are referred to the outpatient cardiology clinics and/or the non-invasive Diagnostic Imaging Department at the local site, have known or suspected CAD and are deemed to clincally require MBF measurements.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terrence Ruddy, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (7):
- Universitaire ziekenhuizen Leuven, Leuven, Belgium
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
- Medizinische Hochschule Hannover, Hanover, Germany
- Nuclear Medicine, Università & Spedali Civili, Brescia, Italy, Brescia, Italy
- Ehime University Hospital, Tōon, Japan
- National Heart Center Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wells RG, Bengel FM, Camoni L, Cerudelli E, Cuddy-Walsh SG, Diekmann J, Han L, Kadoya Y, Kawaguchi N, Keng YJF, Miyagawa M, Ratner H, Teng XF, Ruddy TD. Multicenter Evaluation of the Feasibility of Clinical Implementation of SPECT Myocardial Blood Flow Measurement: Intersite Variability and Imaging Time. Circ Cardiovasc Imaging. 2023 Oct;16(10):e015009. doi: 10.1161/CIRCIMAGING.122.015009. Epub 2023 Oct 6. PMID 37800325

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients will be recruited from those referred to the local site's Diagnostic Imaging Department for SPECT myocardial perfusion imaging (MPI) and who have an intermediate to high pre-test likelihood of disease (Diamond-Forrester criteria ≥ 30%).
Pre-assignment Details: Patients were excluded from the study prior to performing the research imaging if they had PCI or CABG after the consent process. Patients who were found to be pregnant or breastfeeding post consent were also excluded.
Period: Overall Study
Arm/Group | SPECT Imaging With 99mTc-Tetrofosmin
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SPECT Imaging With 99mTc-Tetrofosmin
Number analyzed (Participants) | 35
Age, Continuous [Mean (Full Range); unit: years] | 69 [59 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Suspected or known coronary artery disease [Count of Participants; unit: Participants] | 35

OUTCOME MEASURES:

1. Primary Outcome: Correlation in MBF Between Core Laboratory and Local Site
Description: MBF was measured locally and at a core laboratory using commercially available software. The acquisition protocol was standardized between the local site and core laboratory. a one-day rest-stress protocol was used. Relative perfusion images were obtained after tracer injection. All raw study data were transferred to the core laboratory where processing was independently repeated by one reader to evaluate inter site processing consistency. Perfusion scores were compared with the measured MBF.
Time Frame: The average total amount of time that the patient was assessed for the MBF protocol varied between 71 and 122 minutes.
Population: Myocardial perfusion images were acquired from patients undergoing clinically indicated single photon emission computed tomography myocardial perfusion imaging. Patients were included if they were at least 18 years of age, had a body mass index of less than 40kg/m2, and were of intermediate to high pretest probability of coronary artery disease on a stable medication regimen. All 35 patients scanned were included in the study.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Groups:
- SPECT Imaging With 99mTc-Tetrofosmin: Participants were injected with 42 +/-14 MBq of 99mTc-Tetrofosmin 20 minutes before imaging. dynamic tracer injections were delivered using a syringe pump over a duration of 30 seconds, followed by a 60 second flush. The injection flow rate was 14 mL/min for (7mL tracer, 14 mL flush). List mode data were acquired starting immediately before tracer injection and for a duration of 11 minutes. Relative perfusion images were obtained between 30 and 60 minutes after tracer injection for clinical evaluation. Each site acquired 35 patient data sets which were analyzed as part of the trial. All raw study data was transferred to the core laboratory where processing was independently repeated by one reader to evaluate inter-site processing consistency.
Arm/Group | SPECT Imaging With 99mTc-Tetrofosmin
Number analyzed (Participants) | 35
correlation coefficient | 0.93 [0.87 to 0.97]

2. Secondary Outcome: Impact on Throughput
Description: Additional acquisition time for the MBF acquisition. For each patient study, the time during which the patient was in the camera room for each imaging session was recorded along with the start times for each scan. From this data, the increase in time for MBF protocol compared with the time for a standard myocardial perfusion imaging protocol was determined.
Time Frame: The average total time the patient was in the camera room during the study protocol was 72.28 minutes.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- SPECT Imaging With 99mTc-Tetrofosmin: Participants were injected with 42 +/-14 MBq of 99mTc-Tetrofosmin 20 minutes before imaging. dynamic tracer injections were delivered using a syringe pump over a duration of 30 seconds, followed by a 60 second flush. The injection flow rate was 14 mL/min for (7mL tracer, 14 mL flush). List mode data were acquired starting immediately before tracer injection and for a duration of 11 minutes. Relative perfusion images were obtained between 30 and 60 minutes after tracer injection for clinical evaluation. Each site acquired 35 patient data sets which were analyzed as part of the trial. For each patient study, the time during which the patient was in the camera room for each imaging session was recorded along with the start times for each scan. From this data, the increase in time for MBF protocol compared with the time for a standard myocardial perfusion imaging protocol was determined
Arm/Group | SPECT Imaging With 99mTc-Tetrofosmin
Number analyzed (Participants) | 35
minutes | 72.28 (9.6)

ADVERSE EVENTS:
Time Frame: 12 months, over the course of the whole study.
Arm/Group | SPECT Imaging With 99mTc-Tetrofosmin
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/49/NCT03427749/Prot_SAP_000.pdf